CLINICAL TRIAL: NCT01122342
Title: Vaginal Testosterone Cream For Atrophic Vaginitis in Women Taking Aromatase Inhibitors for Breast Cancer.
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Evaluating outcomes of current subjects pre further enrollment/dose reduction.
Sponsor: University of Vermont (Other)
Responsible Party: Marie Wood, MD, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V0606
Record Dates: First submitted 2010-05-12; First posted 2010-05-13 (Estimated); Last update posted 2010-05-13 (Estimated); Status verified 2010-05

CONDITIONS: Vaginitis; Dyspareunia; Breast Neoplasms
Keywords: Testosterone; Vaginal administration; Aromatase inhibitors
MeSH Terms: conditions — Vaginitis; Dyspareunia; Breast Neoplasms | interventions — Testosterone Propionate; Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaginal Testosterone (Experimental): Daily application of vaginal testosterone for 28 days.
  Interventions: Drug: Testosterone propionate

INTERVENTIONS:
Drug: Testosterone propionate — Testosterone USP micronized powder at a dose of 1mg/gr will be made into a paste with polysorbate 80 NF liquid and will be placed in an emollient cream base. A calibrated applicator will be supplied to measure out doses containing 300mcg of testosterone for daily application. The cream will be applied daily for 28 days. As above if safety and efficacy endpoints are met at this dose a lower dose (150mcg) will be used and if in tun this meets safety and efficacy endpoints a lower dose (75mcg) will be used.
  Other Names: Testosterone cream,; topical testosterone,; vaginal testosterone

SUMMARY:
Atrophic vaginitis is a condition in which the skin lining of the vagina and labia becomes thin and symptoms develop including vaginal itching, vaginal discomfort and dyspareunia. These can significantly affect women's comfort, sexuality and quality of life.

Treatment for this condition includes estrogen given in pill form, commonly known as hormone replacement therapy and local estrogen treatments, such as vaginal estrogen creams and topical vaginal lubricants. Unfortunately, systemic estrogen is contraindicated in many women with breast cancer. Some providers also feel that women who are taking aromatase inhibitors for their breast cancer should also not use local estrogens as several small studies suggest that these treatments might effect estrogen levels and thus might change how effective the aromatase inhibitors are. If these women choose not to use any form of estrogen therapy there symptoms may not be well controlled with other treatments.

The investigators hypothesize that a vaginal testosterone cream might be a safe and effective alternative treatment for these women. This small study is intended to test the hypothesis that testosterone cream will not increase estrogen (estradiol) levels and that it will improve the symptoms of atrophic vaginitis including vaginal dryness, vaginal itching and pain with intercourse.

The investigators will enroll women in the trial who are taking an aromatase inhibitor and have the symptoms mentioned above. They will receive a testosterone cream which will be applied vaginally once a day for 28 days. If good results are found with a prespecified dose of testosterone, a lower dose will be tested in the next group of women enrolled.

DETAILED DESCRIPTION:
Atrophic vaginitis is a condition in which the skin lining of the vagina and labia becomes thin, usually due to a decreased estrogen state - such as menopause. Symptoms of atrophic vaginitis include vaginal itching, vaginal discomfort and dyspareunia and can significantly affect women's comfort, sexuality and quality of life.

Treatment for this condition includes estrogen given in pill form, commonly known as hormone replacement therapy and local estrogen treatments, such as vaginal estrogen creams and topical vaginal lubricants. Unfortunately, systemic estrogen is contraindicated in many women with breast cancer. Some providers also feel that women who are taking aromatase inhibitors for their breast cancer should also not use local estrogens as several small studies suggest that these treatments might effect estrogen levels and thus might change how effective the aromatase inhibitors are. If these women choose not to use any form of estrogen therapy there symptoms may not be well controlled with other treatments.

The investigators hypothesize that a vaginal testosterone cream might be a safe and effective alternative treatment for these women. This small study is intended to test the hypothesis that testosterone cream will not increase estrogen (estradiol) levels and that it will improve the symptoms of atrophic vaginitis including vaginal dryness, vaginal itching and pain with intercourse.

The investigators will enroll women in the trial who are taking an aromatase inhibitor and have the symptoms mentioned above. They will receive a testosterone cream which will be applied vaginally once a day for 28 days. If good results are found with a prespecified dose of testosterone, a lower dose will be tested in the next group of women enrolled.

Objectives:

PRIMARY OBJECTIVE:

1.1. Does topical testosterone cream affect serum estradiol levels in women taking aromatase inhibitors for breast cancer?

SECONDARY OBJECTIVES:

1.2. Can atrophic vaginitis and resultant symptoms of vaginal dryness, itching and dyspareunia in women taking aromatase inhibitors for the treatment of breast cancer be improved with a topical testosterone cream?

1.3. Does topical testosterone cream affect physical findings, pH and cytologic changes in atrophic vaginitis?

Schema:

Intervention - Subjects will apply a testosterone cream to the vaginal area daily for one month (28 days).

Evaluation - Before and after the study intervention participants will have testosterone and high-sensitivity estradiol tested. They will complete a questionnaire on symptoms of atrophic vaginitis and have a gynecologic examination (with visual, speculum, pH and sample of vaginal epithelial cells.)

Endpoints - Serum estradiol levels Improvement in symptoms of atrophic vaginitis, as measured by questionnaire. Atrophic vaginitis as measured by gynecological examination (including pH and cytology to assess maturation index).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed breast cancer (any stage).
* Currently be using an aromatase inhibitor (anastrazole, exemestane or letrozole) for primary or adjuvant breast cancer treatment.
* Must have complaints of vaginal itching, vaginal dryness and/or dyspareunia.
* Not undergoing active chemotherapeutic or radiotherapeutic treatment
* Age >18 years
* Life expectancy of greater than 2 months.
* CALGB (ZUBROD) performance status <3.
* Post-menopausal - defined by absence of menses for at least 12 months and/or an FSH >25. Not post-menopausal as a function of medications intended to suppress ovarian function, such as gonadotropin releasing hormone agonists. Surgically post-menopausal subject eligible.
* The effects of topical testosterone cream on the developing human fetus at the recommended therapeutic dose are unknown. For this study only post-menopausal women are included and all women of child-bearing potential are excluded. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

* Patients who have not recovered from adverse events due to chemotherapeutic agents administered more than 4 weeks earlier.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to testosterone or the emollient delivery cream used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women and women who are breast-feeding are excluded from this study because it is limited to post-menopausal women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-12; Primary Completion 2010-12 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Serum estradiol levels | 28 days
  Will evaluate if serum estradiol levels, measured with a high sensitivity assay, increase in women taking aromatase inhibitors for breast cancer after study intervention of 28 days of vaginal testosterone treatment.

SECONDARY OUTCOMES:
Symptoms of vaginal atrophy | 28 days
  Will evaluate if symptoms of atrophic vaginitis measured on a symptoms questionnaire impove in women taking aromatase inhibitors for breast cancer after study intervention of 28 days of vaginal testosterone treatment.
Clinical signs of vaginal atrophy. | 28 days
  Will evaluate if clinical signs of vaginal atrophy on gynecologic examination decrease in women taking aromatase inhibitors for breast cancer after study intervention of 28 days of vaginal testosterone treatment.
pathologic measures of atrophic vaginitis | 28 days
  Will evaluate if pathologic measures of atrophic vaginitis including maturation index and vaginal pH change in women on aromatase inhibitos for breast cancer after study intervention of 28 days of vaginal testosterone treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina M Witherby, MD, Principal Investigator — Memorial Hospital of Rhode Island, Warren Alpert School od Medicine at Brown University; Hyman Muss, MD, Principal Investigator — University of North Carolina; Marie Wood, MD, Principal Investigator — University of Vermont
Locations (2):
- United States (2):
  - Memorial Hospital of Rhode Island,, Pawtucket, Rhode Island
  - Fletcher Allen Health Care, University of Vermont, Burlington, Vermont